CLINICAL TRIAL: NCT07392281
Title: Efficacy and Mechanisms of Macitentan for Non-Coronary Obstructive Angina
Acronym: MAC-NOCA
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingang Zheng, Head of Department of Cardiology, China-Japan Friendship Hospital, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-351
Record Dates: First submitted 2026-01-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Non-Coronary Obstructive Angina
Keywords: Non-Coronary Obstructive Angina; Coronary microvscular dysfunction; Macitentan; Endothelin-receptor antagonists
MeSH Terms: interventions — macitentan; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taking Macitentan Group (Experimental)
  Interventions: Drug: Macitentan 10 mg tablet, once daily.

INTERVENTIONS:
Drug: Macitentan 10 mg tablet, once daily. — After the patient signed an informed consent form, Macitentan was given as an oral medication (10 mg once daily) for a period of 4 weeks

SUMMARY:
Angina with non-obstructive coronary arteries (ANOCA) is highly prevalent, impairing quality of life and independently associated with cardiovascular events, yet effective treatments are lacking. The endothelin-1 (ET-1)-endothelin receptor (ETR) system is pivotal in ANOCA pathogenesis. Preclinical studies show that ETR blockade or pericyte-specific knockout of ETA receptor improves coronary microcirculatory function in models of myocardial ischemia-reperfusion and diabetes. Clinical evidence indicates ETR antagonists can enhance microvascular endothelial function and myocardial perfusion in ANOCA patients. However, prior studies diagnosed ANOCA based only on symptoms and angiography without precise microvascular functional assessment. Early ETR antagonists also showed frequent adverse effects (e.g., edema, headache), reducing treatment satisfaction. To address this, the investigators will conduct an open-label, single-center, single-arm trial using invasive coronary microcirculatory function testing to accurately phenotype ANOCA and assess microvascular changes. Patients on standard therapy will receive macitentan-a novel ETR antagonist with improved vasodilatory efficacy and safety-to evaluate its effects on coronary microcirculatory function, angina symptoms, and adverse events. Additionally, the investigators will perform multi-omics profiling (proteomics, transcriptomics, metabolomics) on patient blood samples to identify molecular signatures linked to ANOCA subtypes and treatment response, providing evidence for precision intervention strategies in ANOCA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old.
* With typical angina symptoms.
* Excluding obstructive coronary lesions (coronary stenosis ≤50% or FFR ≥0.8) by CAG.
* Coronary microcirculatory function was confirmed via pressure wire-based thermodilution technique.（Patients were classified into subtypes based on coronary microcirculatory function indices: 1) Type I: CFR ≥ 2.5 and IMR < 25; 2) Type II: CFR ≥ 2.5 and IMR ≥ 25; 3) Type III: CFR < 2.5 and IMR < 25; 4) Type IV: CFR < 2.5 and IMR ≥ 25.）
* Sign a written informed consent form.

Exclusion Criteria:

* Pregnant or lactating women.
* History of heart attack within the last 90 days.
* Severe heart disease (e.g., moderate to severe heart failure, severe heart valve disease).
* Severe renal impairment (GFR <30 ml/min/1.73m2).
* Severe liver disease (Child-Pugh class C).
* Moderately severe anaemia (haemoglobin concentration <90 g/L).
* Participation in another drug intervention trial study within the last 90 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in coronary microcirculation function parameters assessed by CFR from baseline to week 4 | the duration of hospital stay, an expected average of 1 week; 4-week follow-up
  Coronary Flow Reserve (CFR): A unitless ratio quantifying maximal coronary blood flow augmentation capacity, measured via thermodilution as the ratio of hyperemic to resting coronary flow. The commonly used cut-off value is 2.0 or 2.5. Increased ratio indicates improved microvascular dilation capacity.
Changes in coronary microcirculation function parameters assessed by IMR from baseline to week 4 | the duration of hospital stay, an expected average of 1 week; 4-week follow-up
  Index of Microcirculatory Resistance (IMR): A pressure-derived metric (units: mmHg·s) assessing microvascular resistance using thermodilution, calculated as distal coronary pressure multiplied by mean transit time during maximal hyperemia. The commonly used cut-off value is 25. Decreased value indicates reduced microvascular resistance.

SECONDARY OUTCOMES:
Change in Score of the Seattle Angina Questionnaire (SAQ) | Endpoint events before administration of macitentan, 1 week and 4 weeks after administration, and 4 weeks after drug withdrawal.
  The Seattle Angina Questionnaire (SAQ) is a 19-item instrument designed to assess the impact of angina on patients' daily lives across five domains: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. Each item is scored on a 0-100 scale, where higher scores indicate fewer symptoms and better quality of life.
Re-hospitalization due to angina pectoris or heart failure, myocardial infarction, and cardiac death. | Endpoint events at 1 week and 4 weeks after administration of macitentan, and 4 weeks after drug withdrawal.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Endpoint events at 1 week and 4 weeks after administration of macitentan, and 4 weeks after drug withdrawal.
  All adverse events such as edema, anemia, headache, dizziness, and hypotension.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China